CLINICAL TRIAL: NCT02849990
Title: A Phase II Neoadjuvant Study of Apalutamide, Abiraterone Acetate, Prednisone, Degarelix and Indomethacin in Men With Localized Prostate Cancer Pre-Prostatectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michael Schweizer, Associate Professor, Division of Medical Oncology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9628; NCI-2016-01027 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9628 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG1716056 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2016-07-25; First posted 2016-07-29 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Stage III Prostate Adenocarcinoma AJCC v7; Stage III Prostate Cancer AJCC v7; Stage IV Prostate Adenocarcinoma AJCC v7; Stage IV Prostate Cancer AJCC v7
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; apalutamide; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Indomethacin; Prednisone; deltacortene; prednylidene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (neoadjuvant chemotherapy) (Experimental): Patients receive androgen receptor antagonist ARN-509 and abiraterone acetate PO daily, prednisone PO BID and indomethacin PO TID. Patients also receive degarelix SC on day 1 and every 4 weeks for 3 doses. Treatment continues for up to 12 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo prostatectomy on day 85.
  Interventions: Drug: Abiraterone Acetate; Drug: Apalutamide; Drug: Degarelix; Drug: Indomethacin; Other: Laboratory Biomarker Analysis; Drug: Prednisone

INTERVENTIONS:
Drug: Abiraterone Acetate — Given PO
  Other Names: CB7630; Zytiga
Drug: Apalutamide — Given PO
  Other Names: ARN 509; ARN-509; ARN509; JNJ 56021927; JNJ-56021927
Drug: Degarelix — Given SC
  Other Names: FE200486; Firmagon
Drug: Indomethacin — Given PO
  Other Names: Indocin; Indometacin
Other: Laboratory Biomarker Analysis — Correlative study
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisonum; Prednitone; Promifen; Servisone; SK-Prednisone

SUMMARY:
This phase II trial studies how well apalutamide, abiraterone acetate, prednisone, degarelix, and indomethacin work in treating patients with prostate cancer that has spread from where it started to nearby tissue or lymph nodes before surgery. Androgen can cause the growth of tumor cells. Hormone therapy using apalutamide, abiraterone acetate, prednisone, degarelix, and indomethacin may fight prostate cancer by lowering the amount of androgen the body makes and/or blocking the use of androgen by the tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The rate of the pathologic complete response (pCR) (i.e. no evidence of residual tumor) as assessed on prostatectomy specimens following 3-months (12 weeks) of neoadjuvant apalutamide, abiraterone acetate, degarelix and indomethacin.

SECONDARY OBJECTIVES:

I. To determine the negative margin rate as assessed on prostatectomy specimens following 3-months (12 weeks) of neoadjuvant apalutamide, abiraterone acetate, degarelix and indomethacin.

II. To determine the rate of near pCR (i.e. =< 5 mm of residual tumor) as assessed on prostatectomy specimens following 3-months (12 weeks) of neoadjuvant apalutamide, abiraterone acetate, degarelix and indomethacin.

III. To determine the rate of pathologic T3 disease as assessed on prostatectomy specimens following 3-months (12 weeks) of neoadjuvant apalutamide, abiraterone acetate, degarelix and indomethacin.

IV. To determine the rate of nodal metastases as assessed on surgical lymph node specimens following 3-months (12 weeks) of neoadjuvant apalutamide, abiraterone acetate, degarelix and indomethacin.

V. To determine the apoptotic index (i.e. percentage of tumor cells undergoing apoptosis) as determined by cleaved caspase-3 immunohistochemistry following 3-months (12 weeks) of neoadjuvant apalutamide, abiraterone acetate, degarelix and indomethacin.

VI. To determine the proportion of men who receive adjuvant radiation therapy within 1-year of prostatectomy.

VII. To determine the biochemical (i.e. prostate-specific antigen [PSA]) progression free survival estimate two years after the last patient has accrued (i.e. confirmed PSA post-radical prostatectomy >= 0.2 ng/mL).

VIII. To determine the overall survival estimate two years after the last patient has accrued.

IX. Safety as assessed by the incidence and severity of adverse events and serious adverse events graded according to the National Cancer Institute - Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

X. Exploratory biomarker assessment.

OUTLINE:

Patients receive apalutamide and abiraterone acetate orally (PO) daily, prednisone PO twice per day (BID) and indomethacin PO three times per day (TID). Patients also receive degarelix subcutaneously (SC) on day 1 and every 4 weeks for 3 doses. Treatment continues for up to 12 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo prostatectomy on day 85.

After completion of study treatment, patients are followed up at 28, 113, 450 and 815 days.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Documented histologically confirmed adenocarcinoma of the prostate
* Willing to undergo prostatectomy as primary treatment for localized prostate cancer
* High risk prostate cancer (per National Comprehensive Cancer Network [NCCN] criteria): Gleason score 8-10 or T3a or PSA > 20 ng/mL or very-high risk prostate cancer (per NCCN criteria): T3b-T4
* Serum testosterone >= 150 ng/dL
* Able to swallow the study drugs whole
* Willing to take abiraterone acetate on an empty stomach (no food should be consumed at least two hours before and for one hour after dosing)
* Agrees to use a condom (even men with vasectomies) and another effective method of birth control if he is having sex with a woman of childbearing potential or agrees to use a condom if he is having sex with a woman who is pregnant while on study drug and for 3 months following the last dose of study drug; must also agree not to donate sperm during the study and for 3 months after receiving the last dose of study drug
* Medications known to lower the seizure threshold (see list under prohibited meds) must be discontinued or substituted at least 4 weeks prior to study entry

Exclusion Criteria:

* Prior local therapy to treat prostate cancer (e.g. radical prostatectomy, radiation therapy, brachytherapy)
* Prior use of apalutamide, abiraterone acetate or degarelix
* Prior or ongoing systemic therapy for prostate cancer including, but not limited to:

  * Hormonal therapy (for example [e.g.] leuprolide, goserelin, triptorelin, degarelix)
  * Cytochrome P450 (CYP)-17 inhibitors (e.g. ketoconazole)
  * Antiandrogens (e.g. bicalutamide, nilutamide)
  * Second generation antiandrogens (e.g. enzalutamide, apalutamide)
  * Immunotherapy (e.g. sipuleucel-T, ipilimumab)
  * Chemotherapy (e.g. docetaxel, cabazitaxel)
* Evidence of serious and/or unstable pre-existing medical, psychiatric or other condition (including laboratory abnormalities) that could interfere with patient safety or provision of informed consent to participate in this study
* Any psychological, familial, sociological, or geographical condition that could potentially interfere with compliance with the study protocol and follow-up schedule
* Absolute neutrophil count [ANC] < 1500/mm^3
* Platelet count < 100,000/mm^3
* Hemoglobin < 9 g/dL
* Total bilirubin > 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >= 2.5 x ULN; Note: in subjects with Gilbert's syndrome, if total bilirubin is > 1.5 x ULN, measure direct and indirect bilirubin and if direct bilirubin is =< 1.5 x ULN, subject may be eligible
* Abnormal kidney function (glomerular filtration rate GFR < 45 mL/min)
* Serum albumin < 3 g/dL
* Serum potassium < 3.5 mmol/L
* Seizure or known condition that may pre-dispose to seizure (e.g. prior stroke within 1 year to randomization, brain arteriovenous malformation, schwannoma, meningioma, or other benign central nervous system [CNS] or meningeal disease which may require treatment with surgery or radiation therapy)
* Severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events (eg, pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias within 6 months prior to randomization
* History of stroke within the last 5-years
* History of gastrointestinal (GI) bleed requiring transfusion
* History of peptic ulcer disease requiring treatment within the last 5-years
* History of asthma that is nonsteroidal anti-inflammatory drug (NSAID)-induced or with asthma that is classified as 'mild-persistent' or worse (based on symptoms occurring more than 2 days per week)
* Uncontrolled hypertension
* Gastrointestinal disorder affecting absorption
* Active infection (eg, human immunodeficiency virus [HIV] or viral hepatitis)
* Any chronic medical condition requiring a higher dose of corticosteroid than 10 mg prednisone/ prednisolone once daily
* Any condition that in the opinion of the investigator, would preclude participation in this study
* Child Pugh class B & C
* Pre-existing viral hepatitis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2020-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schweizer, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Neoadjuvant Chemotherapy)
Started | 22
Completed | 20
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Neoadjuvant Chemotherapy)
Number analyzed (Participants) | 20
Age, Customized [Median (Full Range); unit: years] | 63 [51 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Prostate Specific Antigen (PSA) [Median (Full Range); unit: ng/mL] | 10 [5.6 to 159.4]
Total Gleason score [Median (Full Range); unit: units on a scale] — Gleason score is a pathological assessment based on the architecture of the prostate gland, with Gleason score 1 indicating well differentiated tumors and a score of 5 being the least differentiated. The total Gleason score is the summation of the two most prevalent differentiation patterns observed. Therefore the lowest possible total Gleason score is 2 and the highest is 10. High total Gleason score correlates with poor clinical outcomes.
  units on a scale | 9 [8 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rate as Assessed From Prostatectomy Specimens Following Neoadjuvant Treatment
Description: Pathologic complete response is defined as no evidence of cancer on fully submitted prostatectomy specimens using standard surgical pathology assessments (i.e. H&E assessment will be used for the purpose of defining pathologic complete response per protocol) at 3 months.
Time Frame: At 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Neoadjuvant Chemotherapy)
Number analyzed (Participants) | 20
Participants | 1

2. Secondary Outcome: Apoptotic Index (i.e. Percentage of Tumor Cells Undergoing Apoptosis)
Description: Will be determined by cleaved caspase-3 immunohistochemistry.
Time Frame: At 3 months
Population: Due to limited post-treatment tumor tissue, assessment of apoptotic index is not feasible.
Arm/Group | Treatment (Neoadjuvant Chemotherapy)
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Patients With a Negative Margin After 3 Months of Treatment
Description: The absence of tumor cells at the prostate margin will be assessed using standard pathological practices on prostatectomy specimens (i.e. after 3 months of treatment).
Time Frame: At 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Neoadjuvant Chemotherapy)
Number analyzed (Participants) | 20
Participants
  Negative margins | 13
  Positive margins | 7

4. Secondary Outcome: Overall Survival (OS)
Description: Will will report the number of participants alive at 2-years following enrollment.
Time Frame: At 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Neoadjuvant Chemotherapy)
Number analyzed (Participants) | 20
Participants | 20

5. Secondary Outcome: Number of Patients With a Near Pathologic Complete Response After 3 Months of Treatment
Description: The near pathologic complete response will be defined as =< 5 mm of residual tumor as assessed on prostatectomy specimens after 3 months of treatment.
Time Frame: At 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Neoadjuvant Chemotherapy)
Number analyzed (Participants) | 20
Participants | 6

6. Secondary Outcome: Number of Patients With no Nodal Metastases After 3 Months of Treatment.
Description: The presence of tumor cells within surgically excised lymph nodes will be assessed after 3 months of treament.
Time Frame: At 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Neoadjuvant Chemotherapy)
Number analyzed (Participants) | 20
Participants
  No nodal metastases | 13
  Nodal metastases | 7

7. Secondary Outcome: Number of Patients With Pathologic T3 Disease After 3 Months of Treatment.
Description: The presence of T3 disease (e.g. extraprostatic tumor not invading adjacent structures) will be determine from the prostatectomy specimen after 3 months of treament.
Time Frame: At 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Neoadjuvant Chemotherapy)
Number analyzed (Participants) | 20
Participants | 18

8. Secondary Outcome: Number of Participants Without Biochemical Failure at 2 Years
Description: Prostate-specific antigen progression (i.e. biochemical failure) will be defined per the American Urological Association guidelines (i.e. confirmed prostate-specific antigen post-radical prostatectomy >= 0.2 ng/mL). We will report the number of patients without biochemical failure at 2 years.
Time Frame: At 2 years
Measure: Number; unit: participants
Arm/Group | Treatment (Neoadjuvant Chemotherapy)
Number analyzed (Participants) | 20
participants | 18

9. Secondary Outcome: The Proportion of Men Who Receive Adjuvant Radiation Therapy
Description: Patients that received radiation following prostatetomy
Time Frame: Up to 1 year post prostatectomy
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Neoadjuvant Chemotherapy)
Number analyzed (Participants) | 20
Participants | 7

ADVERSE EVENTS:
Time Frame: Adverse events were assessed for 30 days from the last dose of study drugs. All-cause mortality was assessed up to 2 years.
Arm/Group | Treatment (Neoadjuvant Chemotherapy)
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 22/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Neoadjuvant Chemotherapy) (N=22)
Fatigue (General disorders) | 16
Mood change (General disorders) | 5
Insomnia (General disorders) | 3
Dizziness (General disorders) | 2
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 6
Cognitive Changes (Nervous system disorders) | 11
Headaches (Nervous system disorders) | 2
Balance Problem (Nervous system disorders) | 2
Hot flashes (Endocrine disorders) | 18
Gastrointestinal disorder (General disorders) | 11
Transaminitis (Hepatobiliary disorders) | 4
Injection site reaction (Skin and subcutaneous tissue disorders) | 3
Epistaxis (Blood and lymphatic system disorders) | 3
Hypertension (Vascular disorders) | 9
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/90/NCT02849990/Prot_SAP_000.pdf